CLINICAL TRIAL: NCT03710603
Title: A Phase 3 Study Comparing Daratumumab, VELCADE (Bortezomib), Lenalidomide, and Dexamethasone (D-VRd) vs VELCADE, Lenalidomide, and Dexamethasone (VRd) in Subjects With Previously Untreated Multiple Myeloma Who Are Eligible for High-dose Therapy
Brief Title: Daratumumab, VELCADE (Bortezomib), Lenalidomide and Dexamethasone Compared to VELCADE, Lenalidomide and Dexamethasone in Subjects With Previously Untreated Multiple Myeloma
Acronym: Perseus
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Stichting European Myeloma Network (Network)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Organization: European Myeloma Network B.V. (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMN17/54767414MMY3014
Record Dates: First submitted 2018-10-08; First posted 2018-10-18 (Actual); Results first posted 2024-12-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Bortezomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Velcade Lenalidomide dexamethasone (VRd) (Active Comparator): VRd: subjects will receive VRd for induction and consolidation, followed by lenalidomide (R) maintenance until disease progression or unacceptable toxicity.
  Interventions: Drug: Velcade; Drug: Lenalidomide; Drug: dexamethasone
- Daratumumab + VRd (D-VRd) (Experimental): D-VRd: Subjects will receive D-VRd for induction and consolidation followed by daratumumab and lenalidomide maintenance until disease progression or unacceptable toxicity. Minimal residual disease (MRD)-negative subjects in Arm B will stop therapy with daratumumab after sustained MRD negativity for 12 months and after a minimum of 24 months of maintenance therapy. These subjects will continue lenalidomide maintenance therapy until disease progression or unacceptable toxicity. After stopping daratumumab therapy, subjects with sustained MRD negativity should restart therapy with daratumumab if there is a recurrence of MRD or a confirmed loss of Complete Response (CR) without International Myeloma Working Group (IMWG)-defined disease progression. After reinitiating daratumumab, the subject will continue daratumumab and lenalidomide therapy until disease progression or unacceptable toxicity.
  Interventions: Drug: Daratumumab; Drug: Velcade; Drug: Lenalidomide; Drug: dexamethasone

INTERVENTIONS:
Drug: Daratumumab — Daratumumab will be given at a dose of 1800 mg SC weekly in Cycles 1 and 2, then every 2 weeks in Cycles 3-6. In maintenance Cycles 7+, subjects will receive daratumumab once every 4 weeks until disease progression or unacceptable toxicity. MRD-negative subjects will stop daratumumab after sustained MRD negativity for 12 months & after a min. of 24 months of maintenance. Daratumumab should be restarted at recurrence of MRD or confirmed loss of CR without disease progression.
  Other Names: Velcade (bortezomib); lenalidomide; dexamethasone
  Arms: Daratumumab + VRd (D-VRd)
Drug: Velcade — Bortezomib will be given at a dose of 1.3 mg/m2 SC twice a week (Days 1, 4, 8, and 11) in Cycles 1-6; four 28-day induction cycles (Cycles 1 to 4), and two 28-day consolidation cycles (Cycles 5-6). Subjects will not receive bortezomib after Cycle 6. On treatment days when both bortezomib and daratumumab are administered, bortezomib must be administered after the daratumumab administration.
  Other Names: bortezomib
Drug: Lenalidomide — Lenalidomide will be administered PO at 25 mg on Days 1 to 21 in Cycles 1-6; four 28-day induction cycles and two 28-day consolidation cycles. Following consolidation, subjects will then start maintenance therapy, during which they will receive lenalidomide 10 mg daily PO on Days 1 to 28 (continuously) of each 28-day cycle until disease progression or unacceptable toxicity. After 3 cycles of maintenance therapy, if well tolerated, the lenalidomide dose may be increased to 15 mg daily, at the discretion of the investigator.
Drug: dexamethasone — Dexamethasone will be administered PO at 40 mg daily on Days 1-4 and Days 9-12 of each 28-day cycle during induction and consolidation (Cycles 1-6). On daratumumab administration days, during induction/consolidation, dexamethasone may be administered intravenously 1 hour before the daratumumab administration. On days when daratumumab is not administered, dexamethasone is administered PO. Dexamethasone tablets are to be taken with or immediately after a meal or snack, preferably in the morning.

SUMMARY:
Background of the study: The combination of daratumumab with VRd is anticipated to further improve response rates in patients and may lead to improved long-term outcomes in newly diagnosed patients with multiple myeloma. Given this potential, and based upon the initial safety and efficacy observed in the ongoing Phase 2 Study MMY2004, as well as continued positive results with daratumumab in various disease settings and combination regimens, this Phase 3 study is designed to demonstrate improved outcomes for patients treated with daratumumab+VRd. The Phase 3 study will utilize the subcutaneous (SC) formulation of daratumumab instead of the IV formulation utilized in the Phase 2 study, which may limit additional toxicity to patients treated with the quadruplet regimen.

ELIGIBILITY:
Inclusion Criteria:

1.18 to 70 years of age, inclusive.

2.Monoclonal plasma cells in the bone marrow ≥10% or presence of a biopsy proven plasmacytoma and documented multiple myeloma satisfying at least one of the calcium, renal, anemia, bone (CRAB) criteria or biomarkers of malignancy criteria:

CRAB criteria:

1. Hypercalcemia: serum calcium >0.25 mmol/L (>1 mg/dL) higher than upper limit of normal (ULN) or >2.75 mmol/L (>11 mg/dL)
2. Renal insufficiency: creatinine clearance <40 mL/min or serum creatinine >177 μmol/L (>2 mg/dL)
3. Anemia: hemoglobin >2 g/dL below the lower limit of normal or hemoglobin <10 g/dL
4. Bone lesions: one or more osteolytic lesions on skeletal radiography, CT, or Positron-emission tomography (PET)-CT

Biomarkers of Malignancy:

a. Clonal bone marrow plasma cell percentage ≥60% b. Involved: uninvolved serum free light chain (FLC) ratio ≥100 c. >1 focal lesion on magnetic resonance imaging (MRI) studies

3.Measurable disease as defined by any of the following:

1. Serum monoclonal paraprotein (M-protein) level ≥1.0 g/dL or urine M-protein level ≥200 mg/24 hours; or
2. Light chain multiple myeloma without measurable disease in the serum or the urine: Serum immunoglobulin FLC ≥10 mg/dL and abnormal serum immunoglobulin kappa lambda FLC ratio

   4.Newly diagnosed subjects for whom high-dose therapy and autologous stem cell transplantation (ASCT) is part of the intended treatment plan.

   5.Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2.

   6.Clinical laboratory values meeting the following criteria during the Screening Phase (Screening hematology and chemistry tests should be repeated if done more than 3 days before C1D1):

Adequate bone marrow function:

1. Hemoglobin ≥7.5 g/dL (≥4.65 mmol/L; prior red blood cell (RBC) transfusion or recombinant human erythropoietin use is permitted however transfusions are not permitted within 7 days of randomization to achieve this minimum hemoglobin count);
2. Absolute neutrophil count (ANC) ≥1.0 x 109/L (granulocyte-colony stimulating factor (G-CSF) use is permitted);
3. Platelet count ≥50 x 109/L if bone marrow is >50% involved in myeloma. Otherwise ≥75 x 109/L

Adequate liver function:

1. Aspartate aminotransferase (AST) ≤2.5 x ULN;
2. Alanine aminotransferase (ALT) ≤2.5 x ULN;
3. Total bilirubin ≤1.5 x ULN (except in subjects with congenital bilirubinemia, such as Gilbert syndrome, direct bilirubin ≤1.5 x ULN)

Adequate renal function:

1. Estimated creatinine clearance ≥30 mL/min. Creatinine clearance may be calculated using Cockcroft-Gault, estimated Glomerular filtration rate (eGFR) (Modified Diet in Renal Disease (MDRD)), or Chronic Kidney Disease (CKD)-epi formula
2. Corrected serum calcium ≤13.5 mg/dL (≤3.4 mmol/L); or free ionized calcium ≤6.5 mg/dL (≤1.6 mmol/L)

   7. Female subjects of reproductive childbearing potential must commit to either abstain continuously from heterosexual sexual intercourse or to use 2 methods of reliable birth control simultaneously during the Treatment Period, during any dose interruptions, and for 3 months after the last dose of any component of the treatment regimen. Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study drug. This birth control method must include one highly effective form of contraception (tubal ligation, intrauterine device (IUD), hormonal [birth control pills, injections, hormonal patches, vaginal rings or implants] or partner's vasectomy) and one additional effective contraceptive method (male latex or synthetic condom, diaphragm, or cervical cap). Contraception must begin 4 weeks prior to dosing. Reliable contraception is indicated even where there has been a history of infertility, unless due to hysterectomy or bilateral oophorectomy.

   8. A woman of childbearing potential must have 2 negative serum or urine pregnancy tests at Screening, first within 10 to 14 days prior to dosing and the second within 24 hours prior to dosing.

   9. A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for a period of 3 months after receiving the last dose of any component of the treatment regimen.

   10. Male subjects of reproductive potential who are sexually active with females of reproductive potential must always use a latex or synthetic condom during the study and for 3 months after discontinuing study treatment (even after a successful vasectomy).

   11. Male subjects of reproductive potential must not donate sperm during the study or for 3 months after the last dose of study treatment.

   12. Signed an informed consent form (ICF) (or their legally acceptable representative must sign) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study.

   13. Able to adhere to the prohibitions and restrictions specified in this protocol

Exclusion Criteria:

1. Prior or current systemic therapy or stem cell transplant (SCT) for any plasma cell dyscrasia, with the exception of emergency use of a short course (equivalent of dexamethasone 40 mg/day for a maximum 4 days) of corticosteroids before treatment.
2. Peripheral neuropathy or neuropathic pain Grade 2 or higher, as defined by the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.
3. Prior or concurrent invasive malignancy (other than multiple myeloma) within 5 years of date of randomization (exceptions are adequately treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or breast, or other non-invasive lesion that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence within 3 years).
4. Radiation therapy within 14 days of randomization.
5. Plasmapheresis within 28 days of randomization.
6. Clinical signs of meningeal involvement of multiple myeloma.
7. Chronic obstructive pulmonary disease (COPD) with a Forced Expiratory Volume in 1 second (FEV1) <50% of predicted normal (for subjects ≥65 years old FEV1 <50% or diffusing capacity of the lungs for carbon monoxide [DLCO] <50%)
8. Moderate or severe persistent asthma within the past 2 years, or currently has uncontrolled asthma of any classification. (Note that subjects who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed in the study).
9. Any of the following:

   1. Seropositive for human immunodeficiency virus (HIV)
   2. Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (ie, subjects who are positive for antibodies to hepatitis B core antigen [antiHBc] and/or antibodies to hepatitis B surface antigen [antiHBs]) must be screened using real-time PCR measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (antiHBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by polymerase chain reaction (PCR).
   3. Seropositive for hepatitis C (HCV) (anti-HCV antibody positive or HCV-RNA quantitation positive), except in the setting of a sustained virologic response (SVR), defined as viremia at least 12 weeks after completion of antiviral therapy.
10. Concurrent medical or psychiatric condition or disease (such as but not limited to, systemic amyloidosis, POEMS, active systemic infection, uncontrolled diabetes, acute diffuse infiltrative pulmonary disease) that is likely to interfere with the study procedures or results, or that in the opinion of the investigator, would constitute a hazard for participating in this study.
11. Any of the following:

    1. myocardial infarction within 6 months before randomization, or an unstable or uncontrolled disease/condition related to or affecting cardiac function (eg, unstable angina, congestive heart failure, New York Heart Association Class III-IV)
    2. uncontrolled cardiac arrhythmia or clinically significant electrocardiogram (ECG) abnormalities
    3. screening 12-lead ECG showing a baseline QT interval >470 msec
    4. left ventricular ejection fraction (LVEF) <40% for subjects age 65-70 years old
12. Received a strong CYP3A4 inducer within 5 half-lives prior to randomization
13. Allergy, hypersensitivity, or intolerance to boron or mannitol, corticosteroids, monoclonal antibodies or human proteins, or their excipients (refer to the Investigator's Brochure), or sensitivity to mammalian-derived products or lenalidomide.
14. Not able to comply with the study protocol (eg, because of alcoholism, drug dependency, or psychological disorder). Subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (eg, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.
15. Pregnant, or breast-feeding, or planning to become pregnant while enrolled in this study or within 3 months after the last dose of any component of the treatment regimen. Or, subject is a man who plans to father a child while enrolled in this study or within 3 months after the last dose of any component of the treatment regimen.
16. Major surgery within 2 weeks before randomization or will not have fully recovered from surgery, or has surgery planned during the time the subject is expected to participate in the study. Kyphoplasty or Vertebroplasty is not considered major surgery.
17. Received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 4 weeks before randomization or is currently enrolled in an interventional investigational study.
18. Contraindications to the use of any components of the backbone treatment regimens, per local prescribing information.
19. Gastrointestinal disease that may significantly alter the absorption of oral drugs
20. Vaccination with live attenuated vaccines within 4 weeks of first study agent administration
21. Unable or unwilling to undergo antithrombotic prophylactic treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 709 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2029-11 (Estimated)

CONTACTS AND LOCATIONS:
Locations (13):
- Alfred Hospital, Melbourne, Australia
- University Hospital Leuven, Leuven, Belgium
- University Hospital Ostrava, Ostrava, Czechia
- Odense University Hospital, Odense, Denmark
- CHRU Hôtel Dieu, Nantes, France
- Regional General Hospital Alexandra, Athens, Greece
- Azienda Ospedaliero-Universitaria Ospedali Riuniti Umberto I - G.M. Lancisi - G. Salesi Di Ancona, Ancona, Italy
- Erasmus MC, Rotterdam, Netherlands
- Oslo University Hospital, Oslo, Norway
- Uniwersytet Jagiellonski Collegium Medicum, Krakow, Poland
- Hospital Clinic I Provincial de Barcelona, Barcelona, Spain
- Kantonsspital St. Gallen, Sankt Gallen, Switzerland
- Ankara University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bertamini L, Fokkema C, Rodriguez-Otero P, van Duin M, Terpos E, D'Agostino M, van der Velden VHJ, van de Donk NWCJ, Delforge M, Driessen C, Hajek R, Einsele H, Vangsted A, Vieyra D, Attar R, Sitthi-Amorn A, Carson R, Schjesvold F, Robak P, Beksac M, Spencer A, Broijl A, Cupedo T, Moreau P, Boccadoro M, Sonneveld P. Circulating tumor cells predict myeloma outcomes in patients treated with daratumumab, bortezomib, lenalidomide, and dexamethasone. Blood. 2026 Jan 22;147(4):431-442. doi: 10.1182/blood.2025030113. PMID 41060326
- [Derived] Sanchez Salas JA, Moreno Belmonte MJ, Poveda Garcia A, Ruiz Ruiz E, Soler Espejo E, Cabanas Perianes V, Garcia Hernandez AM. Intestinal Perforation Secondary to Bortezomib-Induced Autonomic Neuropathy. Clin Case Rep. 2025 Apr 1;13(4):e70340. doi: 10.1002/ccr3.70340. eCollection 2025 Apr. PMID 40171013
- [Derived] Sonneveld P, Dimopoulos MA, Boccadoro M, Quach H, Ho PJ, Beksac M, Hulin C, Antonioli E, Leleu X, Mangiacavalli S, Perrot A, Cavo M, Belotti A, Broijl A, Gay F, Mina R, Nijhof IS, van de Donk NWCJ, Katodritou E, Schjesvold F, Sureda Balari A, Rosinol L, Delforge M, Roeloffzen W, Silzle T, Vangsted A, Einsele H, Spencer A, Hajek R, Jurczyszyn A, Lonergan S, Ahmadi T, Liu Y, Wang J, Vieyra D, van Brummelen EMJ, Vanquickelberghe V, Sitthi-Amorn A, de Boer CJ, Carson R, Rodriguez-Otero P, Blade J, Moreau P; PERSEUS Trial Investigators. Daratumumab, Bortezomib, Lenalidomide, and Dexamethasone for Multiple Myeloma. N Engl J Med. 2024 Jan 25;390(4):301-313. doi: 10.1056/NEJMoa2312054. Epub 2023 Dec 12. PMID 38084760
- [Derived] Swan D, Henderson R, McEllistrim C, Naicker SD, Quinn J, Cahill MR, Mykytiv V, Lenihan E, Mulvaney E, Nolan M, Parker I, Natoni A, Lynch K, Ryan AE, Szegezdi E, Krawczyk J, Murphy P, O'Dwyer M. CyBorD-DARA in Newly Diagnosed Transplant-Eligible Multiple Myeloma: Results from the 16-BCNI-001/CTRIAL-IE 16-02 Study Show High Rates of MRD Negativity at End of Treatment. Clin Lymphoma Myeloma Leuk. 2022 Nov;22(11):847-852. doi: 10.1016/j.clml.2022.07.011. Epub 2022 Jul 21. PMID 35985959
- See also: website European Myeloma Network — http://www.myeloma-europe.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Velcade Lenalidomide Dexamethasone (VRd): Arm A: Patients with newly diagnosed multiple myeloma who are eligible for autologous stem cell transplantation were treated with bortezomib, lenalidomide, and dexamethasone for induction and consolidation followed by lenalidomide maintenance in 28-day cycles. After 4 cycles of induction, patients received high dose therapy with autologous stem cell transplantation.
- Daratumumab + VRd (D-VRd): Arm B: Patients with newly diagnosed multiple myeloma who are eligible for autologous stem cell transplantation were treated with subcutaneous daratumumab in combination with bortezomib, lenalidomide, and dexamethasone for induction and consolidation followed by subcutaneous daratumumab in combination with lenalidomide maintenance in 28-day cycles. After 4 cycles of induction, patients received high dose therapy with autologous stem cell transplantation.
Period: Overall Study
Arm/Group | Velcade Lenalidomide Dexamethasone (VRd) | Daratumumab + VRd (D-VRd)
Started | 354 | 355
Completed (Participants that are still on study are listed as "completed") | 295 | 306
Not Completed | 59 | 49
Not completed — Adverse Event | 1 | 0
Not completed — Death | 44 | 34
Not completed — Lost to Follow-up | 3 | 5
Not completed — Withdrawal by Subject | 11 | 10

BASELINE CHARACTERISTICS:
Groups:
- Velcade Lenalidomide Dexamethasone (VRd): Arm A: Patients with newly diagnosed multiple myeloma who are eligible for autologous stem cell transplantation were treated with h bortezomib, lenalidomide, and dexamethasone for induction and consolidation followed by lenalidomide maintenance in 28-day cycles. After 4 cycles of induction, patients received high dose therapy with autologous stem cell transplantation.
- Total: Total of all reporting groups
Arm/Group | Velcade Lenalidomide Dexamethasone (VRd) | Daratumumab + VRd (D-VRd) | Total
Number analyzed (Participants) | 354 | 355 | 709
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (8.12) | 58.7 (7.81) | 58.4 (7.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 144 | 293
  Male | 205 | 211 | 416
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 30 | 50
  Not Hispanic or Latino | 254 | 242 | 496
  Unknown or Not Reported | 80 | 83 | 163
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 4 | 5 | 9
  White | 323 | 330 | 653
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 18 | 12 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 6 | 4 | 10
  Black or African American | 4 | 5 | 9
  Hispanic or Latino | 19 | 28 | 47
  Other | 82 | 83 | 165
  White Non-Hispanic | 243 | 235 | 478
Region of Enrollment [Number; unit: participants]
  Czechia | 4 | 1 | 5
  Switzerland | 5 | 7 | 12
  Spain | 49 | 53 | 102
  Greece | 27 | 32 | 59
  Netherlands | 27 | 30 | 57
  Turkey | 14 | 19 | 33
  Belgium | 10 | 7 | 17
  Norway | 7 | 2 | 9
  Denmark | 9 | 10 | 19
  Poland | 6 | 8 | 14
  Italy | 86 | 64 | 150
  Australia | 38 | 34 | 72
  France | 70 | 83 | 153
  Germany | 2 | 5 | 7
Time Since Initial Diagnosis (months) [Mean (Standard Deviation); unit: months] | 3 (11.41) | 2.2 (4.46) | 2.6 (8.66)
Stage of Disease (ISS) [Count of Participants; unit: Participants] — The International Staging System (ISS) for myeloma was published by the International Myeloma Working Group (a lower stage indicates less progressed disease):
  Stage I: β2-microglobulin (β2M) < 3.5 mg/L, albumin >= 3.5 g/dL Stage II: β2M < 3.5 mg/L and albumin < 3.5 g/dL; or β2M 3.5 mg/L - 5.5 mg/L irrespective of the serum albumin
  Stage III: β2M ≥ 5.5 mg/L.
  Higher stages indicate more advanced disease and/or poorer prognosis.
  Data is the ISS result assessed at the time of randomization.
  Participants
    I | 178 | 186 | 364
    II | 125 | 114 | 239
    III | 50 | 55 | 105
    unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as duration from date of randomization to either progressive disease (PD)/death whichever occurred first. PD was defined as meeting any one of the following criteria: Increase of >= 25 % in level of serum M-protein form lowest response value and absolute increase must be >= 0.5 g/dL; Increase of >=25% in 24-hour urinary light chain excretion (urine M-protein) from lowest response value and absolute increase must be >=200 mg/24 hours; Only in participants without measurable serum and urine M-protein levels; increase of >=25% in difference between involved and uninvolved FLC levels from lowest response value and absolute increase must be > 10 mg/dL; Definite increase in size of existing bone lesions or soft tissue plasmacytomas; Definite development of new bone lesions or soft tissue plasmacytomas; Development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed solely to PC proliferative disorder.
Time Frame: From the date of randomization to either progressive disease or death whichever occurred first, up to a maximum follow-up time of 54.41 months.
Population: Randomized population, intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Velcade Lenalidomide Dexamethasone (VRd) | Daratumumab + VRd (D-VRd)
Number analyzed (Participants) | 354 | 355
Participants | 103 | 50

2. Secondary Outcome: Overall MRD Negativity Rate
Description: Overall MRD-negativity rate was defined as the percentage of participants in the ITT population who achieved both MRD-negativity by NGS (at or below a sensitivity threshold of 10-5) in bone marrow aspirate and a CR or better response at any time after the date of randomization (and prior to disease progression, receipt of subsequent therapy, or both).
Time Frame: From randomization to the clinical cutoff date. Maximum follow up was 54.41 months.
Population: Randomized population, intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Velcade Lenalidomide Dexamethasone (VRd) | Daratumumab + VRd (D-VRd)
Number analyzed (Participants) | 354 | 355
Participants | 168 | 267

3. Secondary Outcome: Percentage of Participants With Overall Response Rate (ORR)
Description: ORR- percentage of participants who achieved partial response (PR) or better (PR, Very Good Partial Response [VGPR], CR or sCR) based on computerized algorithm as per IMWG 2011 criteria. PR -greater than or equal to (>=) 50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >=90% or to <200 mg//24 hours. If serum and urine M-protein are not measurable, a decrease of >=50% in the difference between involved and uninvolved FLC levels is required. A >=50% reduction in the size of soft tissue plasmacytomas is also required; VGPR-serum and urine M-component detectable by immunofixation but not on electrophoresis, or >= 90% reduction in serum M-protein plus urine M-protein <100 mg/24 hours; CR-negative immunofixation on the serum and urine, and disappearance of any soft tissue plasmacytomas, and <5% PCs in bone marrow. sCR- in addition to CR a normal FLC ratio, and absence of clonal PCs by immunohistochemistry or immunofluorescence or 2 to 4-color flow cytometry.
Time Frame: From randomization to the clinical cutoff date. Maximum follow up was 54.41 months
Population: The intent-to-treat (ITT) population included all randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants with response
Arm/Group | Velcade Lenalidomide Dexamethasone (VRd) | Daratumumab + VRd (D-VRd)
Number analyzed (Participants) | 354 | 355
percentage of participants with response | 93.8 [90.7 to 96.1] | 96.6 [94.2 to 98.2]

4. Secondary Outcome: Percentage of Participants With Overall Complete Response (CR) or Better
Description: Percentage of participants achieving CR or better were reported. CR or better rate was defined as the percentage of participants achieving CR or sCR based on the computerized algorithm, according to IMWG response criteria. IMWG 2011 criteria for CR: Negative immunofixation on the serum and urine, and disappearance of any soft tissue plasmacytomas (PCs), and <5% PCs in bone marrow; sCR: CR and normal FLC ratio, absence of clonal PCs by immunohistochemistry, immunofluorescence or 2 to 4 color flow cytometry.
Time Frame: From randomization to the clinical cutoff date. Maximum follow up was 54.41 months
Population: The intent-to-treat (ITT) population included all randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants with response
Arm/Group | Velcade Lenalidomide Dexamethasone (VRd) | Daratumumab + VRd (D-VRd)
Number analyzed (Participants) | 354 | 355
percentage of participants with response | 70.1 [65.0 to 74.8] | 87.9 [84.0 to 91.1]

5. Secondary Outcome: Progression-free Survival on the Next Line of Therapy (PFS2)
Description: Progression-free survival on the next line of therapy (PFS2) is defined as the time from randomization to progression on the next line of treatment or death, whichever comes first.
Time Frame: From randomization to the clinical cutoff date. Maximum follow up was 54.41 months
Reporting Status: Not Posted

6. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS), measured from the date of from randomization to the date the subject's death
Time Frame: From randomization to the clinical cutoff date. Maximum follow up was 54.41 months
Reporting Status: Not Posted

7. Secondary Outcome: Time to Response
Description: Time to response (PR or better), time to CR/sCR are defined as the time from randomization to date of initial response (or initial CR/sCR)
Time Frame: From randomization to the clinical cutoff date. Maximum follow up was 54.41 months
Reporting Status: Not Posted

8. Secondary Outcome: Duration of Response
Description: Duration of response (PR or better), duration of CR, duration of sCR, and duration of MRD-negative status, are calculated from the date of the initial documentation of a response (PR or better), or CR or better, or sCR, or MRD-negative status to the date of the first documented evidence of disease progression, as defined in the IMWG criteria, whichever occurs first.
Time Frame: From randomization to the clinical cutoff date. Maximum follow up was 54.41 months
Reporting Status: Not Posted

9. Secondary Outcome: Pharmacokinetic Concentrations of Daratumumab
Description: Pharmacokinetic concentrations of daratumumab
Time Frame: From randomization to the clinical cutoff date. Maximum follow up was 54.41 months
Reporting Status: Not Posted

10. Secondary Outcome: Determine the Incidence of Anti-daratumumab Antibodies (Immunogenicity) for All Subjects Who Receive at Least 1 Dose of Daratumumab and Determine the Incidence of Anti-rHuPH20 Antibodies
Description: Immunogenicity of daratumumab serum samples will be screened for antibodies binding to daratumumab and serum titer will also be determined from confirmed positive samples using validated immunoassay methods. Other immunogenicity analyses (eg, assessment of neutralizing capabilities) may be performed to further characterize the immune responses that are generated. Plasma samples will be screened for antibodies binding to rHuPH20 and will be assessed in confirmatory and titer assays as necessary
Time Frame: From randomization to the clinical cutoff date. Maximum follow up was 54.41 months
Reporting Status: Not Posted

11. Secondary Outcome: Change in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire 30-item Core Module (EORTC QLQ-C30) Score and the Difference Between-treatment Arms
Description: The EORTC QLQ-C30 is a 30-item questionnaire containing both single and multi-item measures. These include five functional scales (Physical, Role, Cognitive, Emotional, and Social Functioning), three symptom scales (Fatigue, Pain, and Nausea/Vomiting), a Global Health Status/ Quality-of-Life (QoL) scale, and six single items (Constipation, Diarrhea, Insomnia, Dyspnea, Appetite Loss, and Financial Difficulties). The scores ranges from 0-100, a high score for functional scales and for Global Health Status/QoL represent better functioning ability or Health-Related Quality-of-Life (HRQoL), whereas a high score for symptom scales and single items represents significant symptomatology.
Time Frame: From randomization to the clinical cutoff date. Maximum follow up was 54.41 months
Reporting Status: Not Posted

12. Secondary Outcome: Change in EORTC QLQ- 20-item Multiple Myeloma Module (MY-20) Score and the Difference Between-treatment Arms
Description: The EORTC QLQ-MY20 is a supplement to the QLQ-C30 instrument used in subjects with MY. The module comprises 20 questions that address four myeloma-specific HRQoL domains: Disease Symptoms, Side Effects of Treatment, Future Perspective, and Body Image. A high score for Disease Symptoms and Side Effects of Treatment represents a high level of symptomatology or problems, whereas a high score for Future Perspective and Body Image represents better outcomes.
Time Frame: From randomization to the clinical cutoff date. Maximum follow up was 54.41 months
Reporting Status: Not Posted

13. Secondary Outcome: EQ-5D-5L Health Utility Values and the Difference Between-treatment Arms
Description: The EQ-5D-5L is a 5 item questionnaire that assesses 5 domains including mobility, self care, usual activities, pain/discomfort, and anxiety/depression plus a visual analog scale rating "health today"
Time Frame: From randomization to the clinical cutoff date. Maximum follow up was 54.41 months
Reporting Status: Not Posted

14. Secondary Outcome: Stem Cell Yield After Mobilization
Description: Median CD34+ cell yield
Time Frame: From randomization to the clinical cutoff date.
Reporting Status: Not Posted

15. Secondary Outcome: Time to Engraftment Post-ASCT
Description: Time to engraftment post-ASCT defined as absolute neutrophil count (ANC) ≥0.5 x 109/L and platelet count ≥20 x 109/L
Time Frame: From randomization to the clinical cutoff date.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: AEs that started during the treatment until 30 days after the last dose of study treatment. Maximum follow up was 54.41 months.
Description: All-cause mortality is reported for all participants enrolled/randomized in the study (Intent-to-treat population). Serious adverse events and other adverse events are reported for all participants who received at least one dose of study treatment (Safety population).
Arm/Group | Velcade Lenalidomide Dexamethasone (VRd) | Daratumumab + VRd (D-VRd)
All-Cause Mortality (participants affected / at risk) | 44/354 | 34/355
Serious Adverse Events (participants affected / at risk) | 171/347 | 200/351
Other Adverse Events (participants affected / at risk) | 341/347 | 348/351
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Velcade Lenalidomide Dexamethasone (VRd) (N=347) | Daratumumab + VRd (D-VRd) (N=351)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Febrile Bone Marrow Aplasia (Blood and lymphatic system disorders) | 1 | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 16 | 16
Immune Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Thrombotic Microangiopathy (Blood and lymphatic system disorders) | 0 | 1
Acute Coronary Syndrome (Cardiac disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 3
Angina Pectoris (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 2 | 9
Atrial Flutter (Cardiac disorders) | 0 | 1
Cardiac Amyloidosis (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 2 | 0
Cardiac Failure (Cardiac disorders) | 2 | 3
Coronary Artery Disease (Cardiac disorders) | 0 | 3
Left Ventricular Dysfunction (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 4 | 1
Pericardial Effusion (Cardiac disorders) | 1 | 0
Sinus Node Dysfunction (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular Tachycardia (Cardiac disorders) | 0 | 1
Atrial Septal Defect (Congenital, familial and genetic disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 1 | 0
Dacryostenosis Acquired (Eye disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Retinal Detachment (Eye disorders) | 0 | 1
Vision Blurred (Eye disorders) | 0 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1
Anal Fistula (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 2 | 2
Colitis Ulcerative (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 9 | 7
Diverticular Perforation (Gastrointestinal disorders) | 1 | 1
Duodenal Ulcer (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1
Gingival Bleeding (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 2
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Neutropenic Colitis (Gastrointestinal disorders) | 2 | 0
Obstructive Pancreatitis (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 1
Rectal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Asthenia (General disorders) | 0 | 1
Chest Pain (General disorders) | 1 | 0
Chills (General disorders) | 0 | 2
Death (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Gait Disturbance (General disorders) | 0 | 1
Influenza Like Illness (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 16 | 13
Systemic Inflammatory Response Syndrome (General disorders) | 1 | 0
Biliary Dilatation (Hepatobiliary disorders) | 0 | 1
Biliary Obstruction (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 2
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 3
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1
Drug-Induced Liver Injury (Hepatobiliary disorders) | 1 | 1
Hepatic Cytolysis (Hepatobiliary disorders) | 0 | 1
Hepatic Failure (Hepatobiliary disorders) | 0 | 1
Non-Alcoholic Steatohepatitis (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 2 | 0
Abdominal Abscess (Infections and infestations) | 1 | 0
Abscess Neck (Infections and infestations) | 0 | 1
Acute Sinusitis (Infections and infestations) | 0 | 1
Anal Abscess (Infections and infestations) | 1 | 1
Appendicitis (Infections and infestations) | 1 | 0
Appendicitis Perforated (Infections and infestations) | 1 | 1
Bacteraemia (Infections and infestations) | 1 | 1
Bacterial Diarrhoea (Infections and infestations) | 2 | 0
Biliary Tract Infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 3 | 2
Bronchopulmonary Aspergillosis (Infections and infestations) | 1 | 0
Campylobacter Gastroenteritis (Infections and infestations) | 0 | 1
Campylobacter Sepsis (Infections and infestations) | 0 | 1
Chorioretinitis (Infections and infestations) | 0 | 1
Citrobacter Infection (Infections and infestations) | 0 | 1
Clostridium Difficile Colitis (Infections and infestations) | 1 | 1
Clostridium Difficile Infection (Infections and infestations) | 0 | 1
Covid-19 (Infections and infestations) | 6 | 13
Covid-19 Pneumonia (Infections and infestations) | 5 | 11
Cytomegalovirus Enteritis (Infections and infestations) | 0 | 1
Cytomegalovirus Enterocolitis (Infections and infestations) | 1 | 0
Cytomegalovirus Infection Reactivation (Infections and infestations) | 1 | 1
Device Related Infection (Infections and infestations) | 3 | 2
Diverticulitis (Infections and infestations) | 2 | 0
Enterocolitis Viral (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Escherichia Bacteraemia (Infections and infestations) | 0 | 2
Escherichia Peritonitis (Infections and infestations) | 1 | 0
Escherichia Sepsis (Infections and infestations) | 0 | 1
Escherichia Urinary Tract Infection (Infections and infestations) | 1 | 2
Gastroenteritis (Infections and infestations) | 0 | 2
Gastroenteritis Escherichia Coli (Infections and infestations) | 1 | 0
Gastroenteritis Salmonella (Infections and infestations) | 0 | 2
Gastroenteritis Viral (Infections and infestations) | 0 | 2
H1n1 Influenza (Infections and infestations) | 1 | 0
Haemorrhoid Infection (Infections and infestations) | 0 | 1
Hcov-Oc43 Infection (Infections and infestations) | 1 | 0
Hepatitis B Reactivation (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 2
Herpes Zoster Reactivation (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Infestation (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 3
Klebsiella Infection (Infections and infestations) | 2 | 0
Klebsiella Sepsis (Infections and infestations) | 0 | 1
Large Intestine Infection (Infections and infestations) | 1 | 0
Listeria Sepsis (Infections and infestations) | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 3 | 9
Lower Respiratory Tract Infection Bacterial (Infections and infestations) | 0 | 1
Lower Respiratory Tract Infection Viral (Infections and infestations) | 3 | 0
Meningitis Cryptococcal (Infections and infestations) | 1 | 0
Meningitis Listeria (Infections and infestations) | 0 | 1
Mucormycosis (Infections and infestations) | 0 | 1
Neutropenic Sepsis (Infections and infestations) | 0 | 1
Osteomyelitis Salmonella (Infections and infestations) | 1 | 0
Parainfluenzae Virus Infection (Infections and infestations) | 1 | 3
Perirectal Abscess (Infections and infestations) | 1 | 0
Pilonidal Disease (Infections and infestations) | 1 | 0
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 21 | 40
Pneumonia Bacterial (Infections and infestations) | 0 | 2
Pneumonia Cytomegaloviral (Infections and infestations) | 1 | 1
Pneumonia Haemophilus (Infections and infestations) | 0 | 1
Pneumonia Influenzal (Infections and infestations) | 1 | 0
Pneumonia Legionella (Infections and infestations) | 1 | 5
Pneumonia Parainfluenzae Viral (Infections and infestations) | 0 | 1
Pneumonia Pneumococcal (Infections and infestations) | 1 | 3
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 0 | 1
Pneumonia Streptococcal (Infections and infestations) | 0 | 1
Pneumonia Viral (Infections and infestations) | 0 | 1
Post Procedural Sepsis (Infections and infestations) | 0 | 1
Pseudomonal Sepsis (Infections and infestations) | 0 | 1
Pseudomonas Infection (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Respiratory Syncytial Virus Bronchitis (Infections and infestations) | 0 | 1
Respiratory Syncytial Virus Infection (Infections and infestations) | 2 | 2
Respiratory Tract Infection (Infections and infestations) | 1 | 1
Respiratory Tract Infection Viral (Infections and infestations) | 1 | 1
Rhinovirus Infection (Infections and infestations) | 1 | 0
Salmonella Bacteraemia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 9 | 7
Septic Shock (Infections and infestations) | 4 | 3
Sinusitis (Infections and infestations) | 1 | 0
Staphylococcal Abscess (Infections and infestations) | 0 | 1
Staphylococcal Sepsis (Infections and infestations) | 0 | 1
Streptococcal Bacteraemia (Infections and infestations) | 1 | 0
Streptococcal Sepsis (Infections and infestations) | 0 | 1
Subcutaneous Abscess (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 8 | 7
Urinary Tract Infection (Infections and infestations) | 2 | 5
Urosepsis (Infections and infestations) | 1 | 1
Varicella Zoster Virus Infection (Infections and infestations) | 2 | 1
Viral Infection (Infections and infestations) | 1 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 3 | 1
Wound Infection (Infections and infestations) | 0 | 1
Accident (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 3 | 3
Head Injury (Injury, poisoning and procedural complications) | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 1 | 1
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 1
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 3 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 1
Post Procedural Fever (Injury, poisoning and procedural complications) | 0 | 1
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1
Procedural Vomiting (Injury, poisoning and procedural complications) | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 1
Surgical Skin Tear (Injury, poisoning and procedural complications) | 1 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 1
Electrocardiogram Abnormal (Investigations) | 0 | 1
Liver Function Test Abnormal (Investigations) | 0 | 1
Weight Decreased (Investigations) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Diabetic Metabolic Decompensation (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Greater Trochanteric Pain Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis of Jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft Tissue Necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Vertebral Lesion (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute Erythroid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Angioimmunoblastic T-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lentigo Maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Myxofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0
Brain Oedema (Nervous system disorders) | 1 | 0
Brain Stem Stroke (Nervous system disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 3
Chronic Inflammatory Demyelinating Polyradiculoneuropathy (Nervous system disorders) | 0 | 1
Dysaesthesia (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 1
Facial Paralysis (Nervous system disorders) | 0 | 1
Guillain-Barre Syndrome (Nervous system disorders) | 1 | 0
Haemorrhage Intracranial (Nervous system disorders) | 1 | 0
Intensive Care Unit Acquired Weakness (Nervous system disorders) | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 0 | 2
Myelopathy (Nervous system disorders) | 0 | 1
Peripheral Sensorimotor Neuropathy (Nervous system disorders) | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 2
Presyncope (Nervous system disorders) | 1 | 1
Subarachnoid Haemorrhage (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 4
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0
Vith Nerve Paralysis (Nervous system disorders) | 1 | 0
Confusional State (Psychiatric disorders) | 1 | 1
Mania (Psychiatric disorders) | 0 | 1
Psychiatric Decompensation (Psychiatric disorders) | 0 | 1
Psychotic Disorder (Psychiatric disorders) | 1 | 0
Substance-Induced Psychotic Disorder (Psychiatric disorders) | 2 | 0
Acute Kidney Injury (Renal and urinary disorders) | 3 | 1
Bladder Disorder (Renal and urinary disorders) | 0 | 1
Nephrotic Syndrome (Renal and urinary disorders) | 0 | 1
Renal Impairment (Renal and urinary disorders) | 1 | 0
Renal Injury (Renal and urinary disorders) | 1 | 0
Breast Disorder (Reproductive system and breast disorders) | 0 | 1
Cervical Dysplasia (Reproductive system and breast disorders) | 1 | 0
Cystocele (Reproductive system and breast disorders) | 1 | 0
Vaginal Fistula (Reproductive system and breast disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 9
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dermatitis Exfoliative Generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 | 2
Drug Reaction with Eosinophilia and Systemic Symptoms (Skin and subcutaneous tissue disorders) | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Erythrodermic Atopic Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 3 | 2
Embolism (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 2
Jugular Vein Thrombosis (Vascular disorders) | 1 | 1
Orthostatic Hypotension (Vascular disorders) | 1 | 4
Phlebitis (Vascular disorders) | 1 | 0
Subclavian Vein Thrombosis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 1
Vasculitis (Vascular disorders) | 0 | 1
Vena Cava Thrombosis (Vascular disorders) | 1 | 0
Venous Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Velcade Lenalidomide Dexamethasone (VRd) (N=347) | Daratumumab + VRd (D-VRd) (N=351)
Anaemia (Blood and lymphatic system disorders) | 72 | 77
Febrile Neutropenia (Blood and lymphatic system disorders) | 22 | 19
Leukopenia (Blood and lymphatic system disorders) | 14 | 31
Lymphopenia (Blood and lymphatic system disorders) | 9 | 20
Neutropenia (Blood and lymphatic system disorders) | 204 | 241
Thrombocytopenia (Blood and lymphatic system disorders) | 119 | 170
Abdominal Pain (Gastrointestinal disorders) | 37 | 31
Abdominal Pain Upper (Gastrointestinal disorders) | 22 | 33
Constipation (Gastrointestinal disorders) | 118 | 118
Diarrhoea (Gastrointestinal disorders) | 185 | 213
Dyspepsia (Gastrointestinal disorders) | 24 | 30
Nausea (Gastrointestinal disorders) | 58 | 70
Stomatitis (Gastrointestinal disorders) | 30 | 30
Vomiting (Gastrointestinal disorders) | 27 | 38
Asthenia (General disorders) | 89 | 94
Fatigue (General disorders) | 91 | 84
Influenza Like Illness (General disorders) | 32 | 39
Oedema Peripheral (General disorders) | 74 | 72
Pyrexia (General disorders) | 104 | 102
Hypogammaglobulinaemia (Immune system disorders) | 7 | 28
Bronchitis (Infections and infestations) | 37 | 66
Covid-19 (Infections and infestations) | 77 | 115
Gastroenteritis (Infections and infestations) | 13 | 20
Herpes Zoster (Infections and infestations) | 22 | 17
Influenza (Infections and infestations) | 23 | 20
Lower Respiratory Tract Infection (Infections and infestations) | 15 | 19
Nasopharyngitis (Infections and infestations) | 39 | 58
Pneumonia (Infections and infestations) | 21 | 29
Upper Respiratory Tract Infection (Infections and infestations) | 82 | 107
Urinary Tract Infection (Infections and infestations) | 26 | 31
Alanine Aminotransferase Increased (Investigations) | 51 | 57
Aspartate Aminotransferase Increased (Investigations) | 29 | 28
Blood Alkaline Phosphatase Increased (Investigations) | 26 | 18
Gamma-Glutamyltransferase Increased (Investigations) | 27 | 19
Decreased Appetite (Metabolism and nutrition disorders) | 22 | 30
Hyperglycaemia (Metabolism and nutrition disorders) | 15 | 18
Hypocalcaemia (Metabolism and nutrition disorders) | 27 | 24
Hypokalaemia (Metabolism and nutrition disorders) | 43 | 50
Arthralgia (Musculoskeletal and connective tissue disorders) | 69 | 62
Back Pain (Musculoskeletal and connective tissue disorders) | 65 | 78
Bone Pain (Musculoskeletal and connective tissue disorders) | 29 | 29
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 56 | 67
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 16 | 22
Myalgia (Musculoskeletal and connective tissue disorders) | 20 | 29
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 37 | 40
Dizziness (Nervous system disorders) | 34 | 27
Dysgeusia (Nervous system disorders) | 16 | 24
Headache (Nervous system disorders) | 37 | 31
Neuralgia (Nervous system disorders) | 30 | 35
Paraesthesia (Nervous system disorders) | 42 | 46
Peripheral Sensory Neuropathy (Nervous system disorders) | 179 | 188
Tremor (Nervous system disorders) | 18 | 27
Anxiety (Psychiatric disorders) | 18 | 18
Insomnia (Psychiatric disorders) | 61 | 95
Cough (Respiratory, thoracic and mediastinal disorders) | 51 | 85
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 | 37
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 21 | 15
Dry Skin (Skin and subcutaneous tissue disorders) | 13 | 21
Erythema (Skin and subcutaneous tissue disorders) | 18 | 27
Pruritus (Skin and subcutaneous tissue disorders) | 16 | 26
Rash (Skin and subcutaneous tissue disorders) | 94 | 82
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 27 | 26
Hypertension (Vascular disorders) | 21 | 30
Hypotension (Vascular disorders) | 14 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT03710603/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-31): https://cdn.clinicaltrials.gov/large-docs/03/NCT03710603/SAP_001.pdf